CLINICAL TRIAL: NCT00579670
Title: Treatment of Schizophrenic Patients With Geodon; Capsules/Oral Suspension/Solution for Injection (Ziprasidone)
Brief Title: Treatment of Schizophrenic Patients With Ziprasidone
Acronym: TRITON
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1281156
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Results first posted 2010-05-17 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
Keywords: Ziprasidone in patients with schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ziprasidone — Ziprasidone 20mg, 40mg, 60mg, 80mg capsules, hard; Ziprasidone 10 mg/ml oral suspension Ziprasidone 20mg/ml powder and solvent for the reconstitution of solution for injection
  Other Names: Geodon, Zeldox

SUMMARY:
To determine whether ziprasidone provides good efficacy and tolerability in the treatment of schizophrenic Greek patients.

DETAILED DESCRIPTION:
Sampling Method Details: Non-interventional study (subjects chosen by physician in accordance to their usual practice).

ELIGIBILITY:
Inclusion Criteria:

* Usual clinical practice of physician

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Greece (14):
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Chaïdári
  - Pfizer Investigational Site, Corfu
  - Pfizer Investigational Site, Crete
  - Pfizer Investigational Site, Giannitsá
  - Pfizer Investigational Site, Haidari
  - Pfizer Investigational Site, Kalamata
  - Pfizer Investigational Site, Katerini
  - Pfizer Investigational Site, Kozani
  - Pfizer Investigational Site, Lamia
  - Pfizer Investigational Site, Larissa
  - Pfizer Investigational Site, Pátrai
  - Pfizer Investigational Site, Thessaloniki
  - Pfizer Investigational Site, Volos

REFERENCES:
- [Derived] Wang Z, Pang C, Meng Q, Zhang DZ, Hong ZX, He GB, Yang H, Xiang BD, Li X, Jiang TA, Li K, Tang Z, Huang F, Lu M, Yu XL, Cheng ZG, Liu FY, Han ZY, Dou JP, Wu SS, Yu J, Liang P. Laparoscopic hepatectomy versus microwave ablation for multifocal 3-5 cm hepatocellular carcinoma: a multi-centre, real-world study. Int J Surg. 2024 Nov 1;110(11):6911-6921. doi: 10.1097/JS9.0000000000001398. PMID 39699863
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281156&StudyName=Treatment%20of%20schizophrenic%20patients%20with%20Ziprasidone

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The use and dosage of ziprasidone for this Non-interventional Post-Marketing Surveillance study was based on the approved summary of product characteristics (SmPC) document and adjusted solely according to medical and therapeutic necessity.
Groups:
- Ziprasidone < 80 mg: Ziprasidone up to 80 milligrams (mg) per day.
- Ziprasidone 80 mg to < 120 mg: Ziprasidone between 80 mg and < 120 mg per day.
- Ziprasidone 120 mg to < 160 mg: Ziprasidone between 120 mg and < 160 mg per day.
- Ziprasidone >= 160 mg: Ziprasidone 160 mg or greater per day.
- Ziprasidone Unknown: Details are unknown.
Period: Overall Study
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Started | 15 (Full Analysis Set (FAS): at least 1 dose study medication and at least 1 efficacy measurement) | 57 | 88 | 285 | 5
Population: Within SmPC (Started) | 15 (Within summary of product characteristics (SmPC): FAS subjects who received all doses "Within SmPC") | 56 | 83 | 159 | 0 ("Ziprasidone Unknown" reporting group is not applicable to the Within SmPC population)
Population: Within SmPC (Completed) | 13 (Not Completed (DC): Subject died N=1; Adverse Event (AE) N=1) | 55 (DC: Lost to follow-up (LTFU) N=1) | 79 (DC: AE N=1; Lack of efficacy N=1; Other unspecified N=1; Withdrawal by subject N=1) | 147 (DC: AE N=2; Lack of efficacy N=5; LTFU N=3; Other unspecified N=2) | 0
Completed | 13 | 56 | 84 | 263 | 5
Not Completed | 2 | 1 | 4 | 22 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 14 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 4 | 0
Not completed — Other | 0 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown | Total
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5 | 450
Age, Customized [Number; unit: Participants]
  < 18 years | 0 | 0 | 1 | 0 | 0 | 1
  18 years through 44 years | 3 | 22 | 42 | 169 | 2 | 238
  45 years through 64 years | 4 | 19 | 36 | 96 | 2 | 157
  >= 65 years | 8 | 16 | 9 | 20 | 1 | 54
Sex/Gender, Customized [Number; unit: Participants]
  Male | 9 | 35 | 42 | 173 | 3 | 262
  Female | 6 | 22 | 45 | 110 | 2 | 185
  Unspecified | 0 | 0 | 1 | 2 | 0 | 3
Schizophrenia Duration [Mean (Full Range); unit: Years] | 33.9 [0 to 63.1] | 21.4 [0 to 58.5] | 16.9 [0 to 52.4] | 12.8 [0 to 50.3] | 15.6 [0 to 41.4] | 15.4 [0 to 63.1]

OUTCOME MEASURES:

1. Primary Outcome: Summary of Schizophrenia
Description: Stage, symptoms and type of schizophrenia were recorded in addition to demographic and other clinical history data at the Baseline visit. The primary outcome was to assess the participants profile. Some assessments have been included in the Baseline demographics. This outcome presents results for the Summary of Schizophrenia.
Time Frame: Baseline
Population: All subjects randomized to a treatment group were included in the Baseline analysis.
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Stage: First episode | 1 | 5 | 9 | 39 | 0
  Stage: Acute exacerbation | 1 | 2 | 12 | 89 | 2
  Stage: Chronic, stable | 12 | 46 | 54 | 117 | 3
  Stage: Refractory | 1 | 4 | 13 | 40 | 0
  Symptoms: Positive | 2 | 29 | 47 | 191 | 3
  Symptoms: Negative | 6 | 13 | 16 | 49 | 0
  Symptoms: Depressive | 1 | 9 | 9 | 12 | 0
  Symptoms: No predominant symptomatology | 6 | 6 | 16 | 32 | 2
  Type: Catatonic | 1 | 0 | 0 | 7 | 0
  Type: Disorganized | 0 | 0 | 5 | 30 | 0
  Type: Paranoid | 2 | 22 | 43 | 148 | 3
  Type: Residual | 7 | 13 | 14 | 30 | 1
  Type: Undifferentiated | 2 | 5 | 10 | 30 | 0
  Type: Schizoaffective disorder | 3 | 15 | 14 | 35 | 1
  Type: Schizophrenia not otherwise specified (NOS) | 0 | 2 | 2 | 5 | 0

2. Primary Outcome: Summary of Metabolic Risk Factors
Time Frame: Baseline
Population: All subjects randomized to a treatment group were included in this baseline analysis.
Measure: Number; unit: Participants
Groups:
- Ziprasidone Total: Ziprasidone all doses received combined.
Arm/Group | Ziprasidone Total
Number analyzed (Participants) | 450
Participants
  No metabolic risk factors at Baseline | 205
  ≥1 metabolic risk factors at Baseline | 245
  1 metabolic risk factor at Baseline | 133
  2 metabolic risk factors at Baseline | 64
  ≥3 metabolic risk factors at Baseline | 48
  Fasting glucose level (≥110 mg/dL) | 48
  Triglycerides (≥150 mg/dL) | 76
  HDL (men <40 mg/dL; women <50 mg/dL) | 77
  Blood pressure (≥130/85 mm Hg) | 54
  Centrally distributed obesity | 182

3. Primary Outcome: Summary of Most Frequently Used Concomitant Drug Treatments
Description: Most frequently concomitant drug treatments used by >15 participants.
Time Frame: Baseline
Population: All subjects randomized to a treatment group were included in this baseline analysis.
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Akineton | 6 | 11 | 12 | 24 | 0
  Aloperidine | 0 | 6 | 7 | 13 | 0
  Biperiden | 0 | 2 | 5 | 38 | 0
  Clozapine | 3 | 4 | 5 | 4 | 0
  Haloperidol | 1 | 4 | 7 | 45 | 1
  Lorazepam | 0 | 3 | 8 | 33 | 1
  Olanzapine | 0 | 1 | 6 | 20 | 0
  Quetiapine | 0 | 4 | 1 | 10 | 1
  Risperidone | 3 | 7 | 7 | 31 | 1
  Tavor | 1 | 2 | 4 | 9 | 1

4. Secondary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression - Improvement (CGI-I)
Description: CGI-I: 7-point clinician rated scale ranging from 0 (not assessed) to 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 12
Population: The Full Analysis Set (FAS) - all subjects who received at least 1 dose of study medication and have at least 1 efficacy measurement.
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Not assessed | 0 | 1 | 2 | 12 | 0
  Very much improved | 1 | 2 | 7 | 60 | 1
  Much improved | 7 | 18 | 39 | 105 | 2
  Minimally improved | 3 | 33 | 36 | 79 | 1
  No change | 3 | 3 | 3 | 23 | 1
  Minimally worse | 0 | 0 | 0 | 6 | 0

5. Secondary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression of Severity (CGI-S)
Description: CGI-S: 7-point clinician rated scale to assess severity of subject's current illness state; range: 0 (not assessed) to 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected. B = Baseline; F = Final Visit (Week 12)
Time Frame: Baseline, Week 12
Population: FAS; Baseline Visit: 1 subject in the Ziprasidone >=160mg group had missing severity result. Final Visit: 2 subjects (1 subject in the Ziprasidone 120mg to <160mg and 1 subject in the Ziprasidone <80mg group) had missing severity results.
Measure: Number; unit: Participants
Groups:
- Ziprasidone < 80 mg: Ziprasidone up to 80 mg per day.
- Ziprasodone Unknown: Details are unknown.
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasodone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  B - Not assessed | 0 | 0 | 1 | 0 | 0
  F - Not assessed | 0 | 1 | 2 | 12 | 0
  F (only) - Normal, not at all ill | 1 | 0 | 1 | 18 | 0
  B - Borderline mentally ill | 4 | 0 | 2 | 2 | 1
  F - Borderline mentally ill | 3 | 7 | 16 | 47 | 4
  B - Mildly ill | 4 | 11 | 6 | 17 | 2
  F - Mildly ill | 7 | 25 | 33 | 90 | 0
  B - Moderately ill | 6 | 26 | 45 | 80 | 0
  F - Moderately ill | 3 | 17 | 17 | 62 | 0
  B - Markedly ill | 1 | 16 | 24 | 108 | 1
  F - Markedly ill | 0 | 5 | 17 | 40 | 0
  B - Severely ill | 0 | 4 | 10 | 71 | 1
  F - Severely ill | 0 | 2 | 1 | 13 | 1
  B - Among the most extremely ill | 0 | 0 | 0 | 6 | 0
  F - Among the most extremely ill | 0 | 0 | 0 | 3 | 0

6. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) - Positive Subscale
Description: Modified positive subscale: clinician-rated measurement that consists of 30 items, each rated from 1 (absent) to 7 (extreme). Positive subscale (ranging from 4 to 28) taking the sum of the following 4 items: P1, delusions; P2, conceptual disorganization; P3, hallucinatory behavior; and P6, suspiciousness/persecution. Higher scores indicated greater severity of symptoms. The positive subscale total was calculated as the sum of the 4 items in the positive subscale.
Time Frame: Baseline, Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Scores on a scale
  Baseline | 12.9 (4.12) | 14.4 (4.35) | 14.6 (4.82) | 16.6 (5.28) | 12.6 (2.30)
  Final | 10.2 (3.60) | 11.2 (4.35) | 10.5 (4.41) | 10.4 (4.92) | 7.8 (3.03)

7. Secondary Outcome: PANSS - Negative Subscale
Description: Modified negative subscale: assesses negative symptoms associated with schizophrenia. 7 items make up the Negative scale (eg, blunted affect, emotional withdrawal, poor rapport, and passive/apathetic social withdrawal). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total Negative Subscale scores range from 7 to 49. This negative subscale total was calculated as the sum of 4 items in the negative subscale.
Time Frame: Baseline, Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Scores on a scale
  Baseline | 16.7 (4.69) | 16.1 (4.05) | 14.6 (5.30) | 14.7 (5.70) | 12.8 (5.81)
  Final | 14.1 (4.27) | 12.8 (4.67) | 11.3 (4.78) | 10.6 (5.05) | 8.6 (5.18)

8. Secondary Outcome: PANSS - Composite Subscale
Description: The modified composite subscale total was calculated as the difference of the positive subscale total (7 items; total possible score of 49) and the negative subscale total (7 items; total possible score of 49). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The composite subscale total provided an indication of the level of dominance of the symptoms of one subscale over the symptoms of the other subscale. Higher scores indicated greater severity of symptoms.
Time Frame: Baseline, Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Scores on a scale
  Baseline | -3.8 (3.57) | -1.7 (4.86) | 0.0 (5.14) | 1.9 (6.83) | -0.2 (6.14)
  Final | -3.9 (2.82) | -1.5 (3.92) | -0.7 (3.60) | -0.2 (4.57) | -0.8 (2.95)

9. Secondary Outcome: Number of Participants Answering the Question "How Satisfied or Dissatisfied Are You With the Ability of the Medication to Prevent or Treat Your Condition?"
Time Frame: Week 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Extremely Dissatisfied | 0 | 0 | 0 | 1 | 0
  Very Dissatisfied | 0 | 0 | 1 | 5 | 0
  Dissatisfied | 1 | 5 | 3 | 22 | 0
  Somewhat Satisfied | 3 | 15 | 23 | 69 | 1
  Satisfied | 6 | 25 | 40 | 102 | 1
  Very Satisfied | 4 | 11 | 15 | 48 | 3
  Extremely Satisfied | 0 | 0 | 3 | 27 | 0

10. Secondary Outcome: Number of Participants Answering the Question "How Satisfied or Dissatisfied Are You With the Way the Medication Relieves Your Symptoms?"
Time Frame: Week 12
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Extremely Dissatisfied | 0 | 0 | 0 | 1 | 0
  Very Dissatisfied | 0 | 0 | 2 | 6 | 0
  Dissatisfied | 1 | 5 | 1 | 18 | 0
  Somewhat Satisfied | 2 | 14 | 24 | 80 | 1
  Satisfied | 7 | 22 | 38 | 86 | 0
  Very Satisfied | 4 | 14 | 16 | 54 | 2
  Extremely Satisfied | 0 | 1 | 4 | 29 | 2

11. Secondary Outcome: Number of Participants Answering the Question "How Satisfied or Dissatisfied Are You With the Amount of Time it Takes the Medication to Start Working?"
Time Frame: Week 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Extremely Dissatisfied | 0 | 0 | 0 | 2 | 0
  Very Dissatisfied | 0 | 1 | 1 | 4 | 0
  Dissatisfied | 1 | 6 | 6 | 29 | 0
  Somewhat Satisfied | 5 | 21 | 31 | 79 | 0
  Satisfied | 6 | 21 | 32 | 96 | 2
  Very satisfied | 2 | 7 | 12 | 41 | 3
  Extremely satisfied | 0 | 0 | 3 | 23 | 0

12. Secondary Outcome: Number of Participants Answering the Question "As a Result of Taking This Medication, do You Experience Any Side Effects at All?"
Time Frame: Week 12
Measure: Number; unit: Participant
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participant
  Yes | 3 | 11 | 13 | 84 | 1
  No | 11 | 45 | 72 | 189 | 4

13. Secondary Outcome: Number of Participants Answering the Question "How Bothersome Are the Side Effects of the Medication You Take to Treat Your Condition?"
Time Frame: Week 12
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Extremely Bothersome | 0 | 0 | 0 | 1 | 0
  Very Bothersome | 0 | 0 | 1 | 9 | 0
  Somewhat Bothersome | 0 | 8 | 3 | 29 | 0
  A Little Bothersome | 3 | 3 | 7 | 41 | 1
  Not At All Bothersome | 0 | 0 | 2 | 4 | 0

14. Secondary Outcome: Number of Participants Answering the Question "To What Extent do the Side Effects Interfere With Your Physical Health and Ability to Function (ie, Ability to Think Clearly, Stay Awake, Etc)?"
Time Frame: Week 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  A great deal | 0 | 0 | 1 | 6 | 0
  Quite a bit | 0 | 1 | 1 | 11 | 0
  Somewhat | 1 | 4 | 3 | 31 | 0
  Minimally | 2 | 3 | 7 | 28 | 1
  Not at all | 0 | 3 | 1 | 8 | 0

15. Secondary Outcome: Number of Participants Answering the Question "To What Extent do the Side Effects Interfere With Your Mental Function (ie, Ability to Think, Stay Awake, Etc)?"
Time Frame: Week 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  A great deal | 3 | 11 | 13 | 84 | 1
  Quite a bit | 0 | 0 | 0 | 0 | 0
  Somewhat | 0 | 0 | 0 | 0 | 0
  Minimally | 0 | 0 | 0 | 0 | 0
  Not at all | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants Answering the Question "To What Degree Have Medication Side Effects Affected Your Overall Satisfaction With the Medication?"
Time Frame: Week 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  A great deal | 0 | 0 | 1 | 2 | 0
  Quite a bit | 0 | 0 | 1 | 18 | 0
  Somewhat | 1 | 5 | 2 | 26 | 0
  Minimally | 1 | 2 | 4 | 27 | 1
  Not at all | 1 | 4 | 5 | 10 | 0

17. Secondary Outcome: Number of Participants Answering the Question "How Easy or Difficult is it to Use the Medication in Its Current Form?"
Time Frame: Week 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Extremely difficult | 0 | 0 | 0 | 2 | 0
  Very difficult | 0 | 0 | 1 | 2 | 0
  Difficult | 0 | 1 | 3 | 13 | 0
  Somewhat easy | 0 | 9 | 18 | 45 | 0
  Easy | 8 | 25 | 39 | 117 | 3
  Very easy | 4 | 15 | 16 | 71 | 2
  Extremely easy | 2 | 6 | 8 | 22 | 0

18. Secondary Outcome: Number of Participants Answering the Question "How Easy or Difficult is it to Plan When You Will Use the Medication Each Time?"
Time Frame: Week 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Extremely difficult | 0 | 0 | 0 | 0 | 0
  Very difficult | 0 | 0 | 1 | 4 | 0
  Difficult | 1 | 1 | 7 | 25 | 0
  Somewhat easy | 3 | 14 | 21 | 57 | 1
  Easy | 7 | 25 | 37 | 108 | 1
  Very easy | 1 | 7 | 15 | 54 | 3
  Extremely easy | 2 | 9 | 4 | 24 | 0

19. Secondary Outcome: Number of Participants Answering the Question "How Convenient or Inconvenient is it to Take the Medication as Instructed?"
Time Frame: Week 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Extremely inconvenient | 0 | 0 | 0 | 1 | 0
  Very inconvenient | 0 | 0 | 1 | 4 | 0
  Inconvenient | 1 | 4 | 6 | 25 | 0
  Somewhat convenient | 2 | 12 | 30 | 71 | 1
  Convenient | 7 | 26 | 35 | 111 | 1
  Very convenient | 2 | 6 | 7 | 39 | 3
  Extremely convenient | 2 | 8 | 6 | 21 | 0

20. Secondary Outcome: Number of Participants Answering the Question "Overall, How Confident Are You That Taking This Medication is a Good Thing?"
Time Frame: Week 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Not at all confident | 0 | 2 | 2 | 13 | 0
  A little confident | 2 | 10 | 9 | 33 | 1
  Somewhat confident | 6 | 21 | 33 | 88 | 3
  Very confident | 6 | 22 | 34 | 100 | 0
  Extremely confident | 0 | 1 | 7 | 36 | 1

21. Secondary Outcome: Number of Participants Answering the Question "How Certain Are You That the Good Things About Your Medication Outweigh the Bad Things?"
Time Frame: Week 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Not at all certain | 0 | 1 | 2 | 15 | 0
  A little certain | 3 | 13 | 7 | 36 | 0
  Somewhat certain | 6 | 21 | 26 | 81 | 2
  Very certain | 5 | 20 | 44 | 101 | 3
  Extremely certain | 0 | 1 | 6 | 39 | 0

22. Secondary Outcome: Number of Participants Answering the Question "Taking All Things Into Account, How Satisfied or Dissatisfied Are You With This Medication?"
Time Frame: Week 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Extremely dissatisfied | 0 | 0 | 0 | 2 | 0
  Very dissatisfied | 0 | 0 | 0 | 6 | 0
  Dissatisfied | 1 | 5 | 3 | 17 | 0
  Somewhat satisfied | 1 | 19 | 16 | 64 | 1
  Satisfied | 7 | 17 | 37 | 89 | 1
  Very satisfied | 5 | 15 | 23 | 61 | 2
  Extremely satisfied | 0 | 0 | 5 | 32 | 1

23. Other Pre Specified Outcome: Number of Participants Continuing Treatment With Ziprasidone Following Completion of the Observation Period
Time Frame: Week 12
Population: FAS. Four subjects did not answer the question of continuation of treatment.
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
Participants
  Yes | 13 | 56 | 83 | 245 | 4
  No | 2 | 1 | 4 | 38 | 0

24. Secondary Outcome: Percent Change From Baseline to Final Visit in Body Weight
Time Frame: Baseline, Week 12
Population: Safety population = all subjects who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >= 160 mg | Ziprasidone Unknown
Number analyzed (Participants) | 15 | 57 | 88 | 285 | 5
percent change | 1.2 (5.79) | -0.2 (3.67) | -1.0 (3.08) | 0.1 (4.70) | -1.0 (2.05)

25. Post Hoc Outcome: Number of Participants With Categorical Scores on Clinical Global Impression - Improvement (CGI-I): Within Summary of Product Characteristics Population (SmPC)
Description: as for outcome 4
Time Frame: Week 12
Population: Within SmPC population: participants in FAS population who received all doses within SmPC. Within SmPC defined as all PO doses up to and including 160 mg per day and all IM doses up to and including 40 mg per day.
Measure: Number; unit: Participants
Groups:
- Ziprasidone < 80 mg: Ziprasidone up to 80 mg orally (PO) per day or up to 40 mg intramuscularly (IM) per day.
- Ziprasidone 80 mg to < 120 mg: Ziprasidone between 80 mg and < 120 mg PO per day.
- Ziprasidone 120 mg to < 160 mg: Ziprasidone between 120 mg and < 160 mg PO per day.
- Ziprasidone = 160 mg: Ziprasidone 160 mg PO per day.
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 15 | 56 | 83 | 159
Participants
  Not assessed | 0 | 1 | 2 | 6
  Very much improved | 1 | 2 | 6 | 22
  Much improved | 7 | 17 | 39 | 62
  Minimally improved | 3 | 33 | 32 | 52
  No change | 3 | 3 | 3 | 14
  Minimally worse | 0 | 0 | 0 | 3

26. Post Hoc Outcome: Number of Participants With Categorical Scores on Clinical Global Impression of Severity (CGI-S): Within SmPC
Description: as for outcome 5
Time Frame: Baseline, Week 12
Population: Within SmPC
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 15 | 56 | 83 | 159
Participants
  B - Not assessed | 0 | 0 | 1 | 0
  F - Not assessed | 0 | 1 | 2 | 6
  F (only) - Normal, not at all ill | 1 | 0 | 1 | 6
  B - Borderline mentally ill | 4 | 0 | 2 | 1
  F - Borderline mentally ill | 3 | 7 | 14 | 24
  B - Mildly ill | 4 | 11 | 5 | 10
  F - Mildly ill | 7 | 24 | 31 | 53
  B - Moderately ill | 6 | 25 | 41 | 53
  F - Moderately ill | 3 | 17 | 16 | 38
  B - Markedly ill | 1 | 16 | 24 | 59
  F - Markedly ill | 0 | 5 | 17 | 22
  B - Severely ill | 0 | 4 | 10 | 33
  F - Severely ill | 0 | 2 | 1 | 8
  B - Among the most extremely ill | 0 | 0 | 0 | 2
  F - Among the most extremely ill | 0 | 0 | 0 | 2

27. Post Hoc Outcome: Positive and Negative Syndrome Scale (PANSS) - Positive Subscale: Within SmPC
Description: as for outcome 6
Time Frame: Baseline, Week 12
Population: Within SmPC; N=participants with evaluable data at observation
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 15 | 56 | 82 | 158
Scores on a scale
  Baseline | 12.9 (4.12) | 14.5 (4.37) | 14.8 (4.85) | 15.3 (5.27)
  Final | 10.2 (3.60) | 11.3 (4.38) | 10.7 (4.47) | 10.0 (4.51)

28. Post Hoc Outcome: PANSS - Negative Subscale: Within SmPC
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: Within SmPC; N=participants with evaluable data at observation
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 15 | 55 | 82 | 157
Scores on a scale
  Baseline | 16.7 (4.69) | 16.0 (4.06) | 14.8 (5.22) | 14.5 (5.91)
  Final | 14.1 (4.27) | 12.7 (4.71) | 11.4 (4.76) | 11.1 (5.33)

29. Post Hoc Outcome: PANSS - Composite Subscale: Within SmPC
Description: as for outcome 8
Time Frame: Baseline, Week 12
Population: Within SmPC; N=participants with evaluable data at observation
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 15 | 55 | 82 | 157
Scores on a scale
  Baseline | -3.8 (3.57) | -1.5 (4.80) | 0.0 (5.09) | 0.7 (7.32)
  Final | -3.9 (2.82) | -1.5 (3.91) | -0.6 (3.58) | -1.1 (4.61)

30. Post Hoc Outcome: Number of Participants Answering the Question "How Satisfied or Dissatisfied Are You With the Ability of the Medication to Prevent or Treat Your Condition?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 14 | 55 | 80 | 153
Participants
  Extremely Dissatisfied | 0 | 0 | 0 | 0
  Very Dissatisfied | 0 | 0 | 1 | 3
  Dissatisfied | 1 | 5 | 3 | 12
  Somewhat Satisfied | 3 | 15 | 23 | 43
  Satisfied | 6 | 24 | 36 | 56
  Very Satisfied | 4 | 11 | 14 | 30
  Extremely Satisfied | 0 | 0 | 3 | 9

31. Post Hoc Outcome: Number of Participants Answering the Question "How Satisfied or Dissatisfied Are You With the Way the Medication Relieves Your Symptoms?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 14 | 55 | 80 | 153
Participants
  Extremely Dissatisfied | 0 | 0 | 0 | 0
  Very Dissatisfied | 0 | 0 | 2 | 3
  Dissatisfied | 1 | 5 | 1 | 11
  Somewhat Satisfied | 2 | 14 | 24 | 48
  Satisfied | 7 | 21 | 34 | 48
  Very Satisfied | 4 | 14 | 15 | 34
  Extremely Satisfied | 0 | 1 | 4 | 9

32. Post Hoc Outcome: Number of Participants Answering the Question "How Satisfied or Dissatisfied Are You With the Amount of Time it Takes the Medication to Start Working?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 14 | 55 | 80 | 153
Participants
  Extremely Dissatisfied | 0 | 0 | 0 | 0
  Very Dissatisfied | 0 | 1 | 1 | 3
  Dissatisfied | 1 | 6 | 6 | 17
  Somewhat Satisfied | 5 | 20 | 30 | 42
  Satisfied | 6 | 21 | 28 | 58
  Very satisfied | 2 | 7 | 12 | 26
  Extremely satisfied | 0 | 0 | 3 | 7

33. Post Hoc Outcome: Number of Participants Answering the Question "As a Result of Taking This Medication, do You Experience Any Side Effects at All?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participant
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 14 | 55 | 80 | 152
Participant
  Yes | 3 | 11 | 13 | 41
  No | 11 | 44 | 67 | 111

34. Post Hoc Outcome: Number of Participants Answering the Question "How Bothersome Are the Side Effects of the Medication You Take to Treat Your Condition?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 3 | 11 | 13 | 41
Participants
  Extremely Bothersome | 0 | 0 | 0 | 0
  Very Bothersome | 0 | 0 | 1 | 4
  Somewhat Bothersome | 0 | 8 | 3 | 18
  A Little Bothersome | 3 | 3 | 7 | 18
  Not At All Bothersome | 0 | 0 | 2 | 1

35. Post Hoc Outcome: Number of Participants Answering the Question "To What Extent do the Side Effects Interfere With Your Physical Health and Ability to Function (ie, Ability to Think Clearly, Stay Awake, Etc)?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 3 | 11 | 13 | 41
Participants
  A great deal | 0 | 0 | 1 | 1
  Quite a bit | 0 | 1 | 1 | 7
  Somewhat | 1 | 4 | 3 | 18
  Minimally | 2 | 3 | 7 | 12
  Not at all | 0 | 3 | 1 | 3

36. Post Hoc Outcome: Number of Participants Answering the Question "To What Extent do the Side Effects Interfere With Your Mental Function (ie, Ability to Think, Stay Awake, Etc)?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 3 | 11 | 13 | 41
Participants
  A great deal | 3 | 11 | 13 | 41
  Quite a bit | 0 | 0 | 0 | 0
  Somewhat | 0 | 0 | 0 | 0
  Minimally | 0 | 0 | 0 | 0
  Not at all | 0 | 0 | 0 | 0

37. Post Hoc Outcome: Number of Participants Answering the Question "To What Degree Have Medication Side Effects Affected Your Overall Satisfaction With the Medication?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 3 | 11 | 13 | 41
Participants
  A great deal | 0 | 0 | 1 | 2
  Quite a bit | 0 | 0 | 1 | 8
  Somewhat | 1 | 5 | 2 | 15
  Minimally | 1 | 2 | 4 | 12
  Not at all | 1 | 4 | 5 | 4

38. Post Hoc Outcome: Number of Participants Answering the Question "How Easy or Difficult is it to Use the Medication in Its Current Form?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 14 | 55 | 80 | 152
Participants
  Extremely difficult | 0 | 0 | 0 | 2
  Very difficult | 0 | 0 | 1 | 1
  Difficult | 0 | 1 | 3 | 9
  Somewhat easy | 0 | 9 | 17 | 22
  Easy | 8 | 24 | 36 | 65
  Very easy | 4 | 15 | 15 | 44
  Extremely easy | 2 | 6 | 8 | 9

39. Post Hoc Outcome: Number of Participants Answering the Question "How Easy or Difficult is it to Plan When You Will Use the Medication Each Time?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 14 | 55 | 80 | 152
Participants
  Extremely difficult | 0 | 0 | 0 | 0
  Very difficult | 0 | 0 | 1 | 3
  Difficult | 1 | 1 | 6 | 16
  Somewhat easy | 3 | 14 | 20 | 32
  Easy | 7 | 24 | 35 | 60
  Very easy | 1 | 7 | 14 | 30
  Extremely easy | 2 | 9 | 4 | 11

40. Post Hoc Outcome: Number of Participants Answering the Question "How Convenient or Inconvenient is it to Take the Medication as Instructed?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 14 | 55 | 80 | 152
Participants
  Extremely inconvenient | 0 | 0 | 0 | 1
  Very inconvenient | 0 | 0 | 1 | 2
  Inconvenient | 1 | 4 | 6 | 13
  Somewhat convenient | 2 | 12 | 28 | 38
  Convenient | 7 | 25 | 33 | 67
  Very convenient | 2 | 6 | 6 | 20
  Extremely convenient | 2 | 8 | 6 | 11

41. Post Hoc Outcome: Number of Participants Answering the Question "Overall, How Confident Are You That Taking This Medication is a Good Thing?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 14 | 55 | 80 | 152
Participants
  Not at all confident | 0 | 2 | 2 | 7
  A little confident | 2 | 10 | 9 | 23
  Somewhat confident | 6 | 20 | 32 | 49
  Very confident | 6 | 22 | 30 | 57
  Extremely confident | 0 | 1 | 7 | 16

42. Post Hoc Outcome: Number of Participants Answering the Question "How Certain Are You That the Good Things About Your Medication Outweigh the Bad Things?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 14 | 55 | 80 | 152
Participants
  Not at all certain | 0 | 1 | 2 | 8
  A little certain | 3 | 13 | 7 | 23
  Somewhat certain | 6 | 21 | 26 | 47
  Very certain | 5 | 19 | 39 | 56
  Extremely certain | 0 | 1 | 6 | 18

43. Post Hoc Outcome: Number of Participants Answering the Question "Taking All Things Into Account, How Satisfied or Dissatisfied Are You With This Medication?": Within SmPC
Time Frame: Week 12
Population: Within SmPC; N=participants with evaluable data for specified question at observation
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 14 | 55 | 79 | 152
Participants
  Extremely dissatisfied | 0 | 0 | 0 | 1
  Very dissatisfied | 0 | 0 | 0 | 2
  Dissatisfied | 1 | 5 | 3 | 10
  Somewhat satisfied | 1 | 19 | 16 | 43
  Satisfied | 7 | 16 | 33 | 47
  Very satisfied | 5 | 15 | 22 | 37
  Extremely satisfied | 0 | 0 | 5 | 12

44. Post Hoc Outcome: Percent Change From Baseline to Final Visit in Body Weight: Within SmPC
Time Frame: Baseline, Week 12
Population: Within SmPC
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 15 | 56 | 83 | 159
percent change | 1.2 (5.79) | -0.2 (3.67) | -1.1 (2.75) | -0.0 (4.31)

45. Post Hoc Outcome: Number of Participants Continuing Treatment With Ziprasidone Following Completion of the Observation Period: Within SmPC
Time Frame: Week 12
Population: Within SmPC
Measure: Number; unit: Participants
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone = 160 mg
Number analyzed (Participants) | 15 | 56 | 83 | 159
Participants
  Yes | 13 | 55 | 78 | 136
  No | 2 | 1 | 4 | 23

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Ziprasidone >=160 mg: Ziprasidone 160 mg or greater per day.
- Within SmPC Ziprasidone < 80 mg: Within SmPC < 80 mg per day; defined as all participants in the FAS population who had PO doses up to 80 mg per day and all IM doses up to and including 40 mg per day.
- Within SmPC Ziprasidone 80 to < 120 mg: Within SmPC Ziprasidone 80 to < 120 mg; defined as all participants in the FAS population who had PO doses between 80 mg and < 120 mg per day.
- Within SmPC Ziprasidone 120 to < 160 mg: Within SmPC Ziprasidone 120 to < 160 mg; defined as all participants in the FAS population who had PO doses between 120 mg and < 160 mg per day.
- Within SmPC Ziprasidone = 160 mg: Within SmPC Ziprasidone = 160 mg; defined as all participants in the FAS population who had PO doses = 160 mg per day.
- Above SmPC Ziprasidone > 160 mg: Above SmPC Ziprasidone > 160 mg per day; defined as all participants in FAS population who received at least 1 PO dose above 160 mg per day or any IM dose above 40 mg per day or with an unknown dose or formulation.
Arm/Group | Ziprasidone < 80 mg | Ziprasidone 80 mg to < 120 mg | Ziprasidone 120 mg to < 160 mg | Ziprasidone >=160 mg | Ziprasidone Unknown | Within SmPC Ziprasidone < 80 mg | Within SmPC Ziprasidone 80 to < 120 mg | Within SmPC Ziprasidone 120 to < 160 mg | Within SmPC Ziprasidone = 160 mg | Above SmPC Ziprasidone > 160 mg
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/57 | 0/88 | 1/285 | 0/5 | 1/15 | 0/56 | 0/83 | 1/159 | 0/128
Other Adverse Events (participants affected / at risk) | 1/15 | 0/57 | 9/88 | 34/285 | 1/5 | 1/15 | 0/56 | 9/83 | 19/159 | 17/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone < 80 mg (N=15) | Ziprasidone 80 mg to < 120 mg (N=57) | Ziprasidone 120 mg to < 160 mg (N=88) | Ziprasidone >=160 mg (N=285) | Ziprasidone Unknown (N=5) | Within SmPC Ziprasidone < 80 mg (N=15) | Within SmPC Ziprasidone 80 to < 120 mg (N=56) | Within SmPC Ziprasidone 120 to < 160 mg (N=83) | Within SmPC Ziprasidone = 160 mg (N=159) | Above SmPC Ziprasidone > 160 mg (N=128)
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ziprasidone < 80 mg (N=15) | Ziprasidone 80 mg to < 120 mg (N=57) | Ziprasidone 120 mg to < 160 mg (N=88) | Ziprasidone >=160 mg (N=285) | Ziprasidone Unknown (N=5) | Within SmPC Ziprasidone < 80 mg (N=15) | Within SmPC Ziprasidone 80 to < 120 mg (N=56) | Within SmPC Ziprasidone 120 to < 160 mg (N=83) | Within SmPC Ziprasidone = 160 mg (N=159) | Above SmPC Ziprasidone > 160 mg (N=128)
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 9 | 0 | 0 | 0 | 2 | 3 | 6
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 3 | 4
Somnolence (Nervous system disorders) | 0 | 0 | 4 | 15 | 1 | 0 | 0 | 4 | 9 | 6
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 4 | 0 | 1 | 0 | 1 | 3 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 0 | 1 | 3

LIMITATIONS AND CAVEATS:
Additional descriptive tables were identified as required after review of the originally planned study tables; many subjects included in the tables had received ziprasidone doses above those specified in the summary of product characteristics (SmPC).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other